CLINICAL TRIAL: NCT00395993
Title: Comparison of the Safety and Efficacy of Intravenous Iron vs Oral Iron in the Treatment of Anemia Secondary to Heavy Uterine Bleeding
Brief Title: Comparison of the Safety and Efficacy of Intravenous Iron Versus Oral Iron in the Treatment of Anemia Secondary to Heavy Uterine Bleeding
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1VIT04002/003
Record Dates: First submitted 2006-11-02; First posted 2006-11-06 (Estimated); Results first posted 2013-11-18 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-01

CONDITIONS: Anemia
Keywords: anemia; heavy uterine bleeding; menorrhagia; Anemia secondary to heavy uterine bleeding
MeSH Terms: conditions — Anemia; Menorrhagia | interventions — ferric carboxymaltose; Iron-Dextran Complex; Iron

ARMS (2):
- Ferric Carboxymaltose (FCM) (Experimental): Maximum of 1,000 mg of iron as IV FCM given at weekly intervals until the individual's calculated cumulative dose has been reached or a maximum of 2,500 mg has been administered
  Interventions: Drug: Ferric Carboxymaltose (FCM)
- Ferrous Sulfate tablets (Active Comparator): 325 mg tablets TID on Days 0 through Day 42
  Interventions: Drug: Ferrous Sulfate tablets

INTERVENTIONS:
Drug: Ferric Carboxymaltose (FCM) — Maximum of 1,000 mg of iron as IV FCM given at weekly intervals until the individual's calculated cumulative dose has been reached or a maximum of 2,500 mg has been administered
  Arms: Ferric Carboxymaltose (FCM)
Drug: Ferrous Sulfate tablets — 325 mg tablets TID on Days 0 through Day 42
  Other Names: Oral Iron Tablets
  Arms: Ferrous Sulfate tablets

SUMMARY:
This study compares of the safety and efficacy of intravenous iron vs oral iron in the treatment of anemia secondary to heavy uterine bleeding

DETAILED DESCRIPTION:
This is an open-label, randomized, Phase III, active-control, study of the efficacy and safety of IV iron vs oral iron in patients with anemia secondary to heavy uterine bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects >/= 18 years of age
* History of Heavy uterine bleeding
* Hgb </= 11
* Practicing acceptable birth control
* Demonstrate ability to understand and comply with protocol

Exclusion Criteria:

* Known Hypersensitivity to oral or IV iron
* Anemia other than iron deficiency anemia
* Iron storage disorders
* Initiation of treatment that may effect degree of heavy uterine bleeding
* Anticipated need for surgery
* Severe psychiatric disorder
* Active infection
* Positive Pregnancy test
* Known Hep B or C or Active Hepatitis
* Received investigational Drug within 30 days
* Alcohol or drug abuse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Actual)
Dates: Start 2005-05; Primary Completion 2006-04 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Luitpold Pharmaceuticals, Inc., Norristown, Pennsylvania, United States

REFERENCES:
- [Result] Gordon S, Hadley PE, Van Wyck DB, Mangione A. Ferric Carboxymaltose, a New IV Iron Agent for Iron Deficiency Anemia in Heavy Uterine Bleeding. Society for the Advancement of Blood Management 6th Annual Meeting 2007.
- [Result] Gordon S, Hadley PE, Van Wyck DB, Mangione A. Iron Carboxymaltose, a New Intravenous Iron Agent for Iron Deficiency Anemia in Heavy Uterine Bleeding. American College of Obstetricians & Gynecologists: 108S 2007.
- [Result] Morrison J, Patel ST, Watson W, Zaidi QR, Mangione A, Goss TF. Assessment of the prevalence and impact of anemia on women hospitalized for gynecologic conditions associated with heavy uterine bleeding. J Reprod Med. 2008 May;53(5):323-30. PMID 18567277
- [Result] James AH, Patel ST, Watson W, Zaidi QR, Mangione A, Goss TF. An assessment of medical resource utilization and hospitalization cost associated with a diagnosis of anemia in women with obstetrical bleeding in the United States. J Womens Health (Larchmt). 2008 Oct;17(8):1279-84. doi: 10.1089/jwh.2007.0605. PMID 18752459
- [Derived] Van Wyck DB, Mangione A, Morrison J, Hadley PE, Jehle JA, Goodnough LT. Large-dose intravenous ferric carboxymaltose injection for iron deficiency anemia in heavy uterine bleeding: a randomized, controlled trial. Transfusion. 2009 Dec;49(12):2719-28. doi: 10.1111/j.1537-2995.2009.02327.x. Epub 2009 Jul 22. PMID 19682342

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hospitals and medical clinics
Groups:
- Oral Iron Tablets: 325 mg tablets TID on Days 0 through Day 42
Period: Overall Study
Arm/Group | Ferric Carboxymaltose (FCM) | Oral Iron Tablets
Started | 246 | 231
Completed | 211 | 212
Not Completed | 35 | 19

BASELINE CHARACTERISTICS:
Population: 16 of the 246 subjects randomized to FCM were discontinued prior to dosing and 5 of the 231 subjects randomized to oral iron were discontinued prior to dosing.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ferric Carboxymaltose (FCM) | Oral Iron Tablets | Total
Number analyzed (Participants) | 230 | 226 | 456
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 0 | 2
  Between 18 and 65 years | 228 | 226 | 454
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (7.49) | 39.5 (7.63) | 39.1 (7.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 230 | 226 | 456
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 230 | 226 | 456

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Achieving 'Clinical Success'. Clinical Success is Defined as an Increase in Hemoglobin of ≥ 2.0 g/dL
Time Frame: Any time between baseline and the end of study or time to intervention
Population: Modified Intent-to-Treat Population defined as subjects from the Safety Population who received at least 1 dose of study medication, had average baseline hemoglobin, TSAT, and ferritin levels, had heavy uterine bleeding, and had at least 1 post-baseline hemoglobin assessment.
Measure: Number; unit: participants
Arm/Group | Ferric Carboxymaltose (FCM) | Oral Iron Tablets
Number analyzed (Participants) | 228 | 225
participants | 187 | 139

ADVERSE EVENTS:
Time Frame: 11 months
Arm/Group | Ferric Carboxymaltose (FCM) | Oral Iron Tablets
Serious Adverse Events (participants affected / at risk) | 3/230 | 3/226
Other Adverse Events (participants affected / at risk) | 120/230 | 133/226
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ferric Carboxymaltose (FCM) (N=230) | Oral Iron Tablets (N=226)
Uterine hemorrhage (Reproductive system and breast disorders) | 1 | 1
Transient ischemic attack (Nervous system disorders) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chest pain (General disorders) | 1 | 0
Pelvic inflammatory disease (Infections and infestations) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ferric Carboxymaltose (FCM) (N=230) | Oral Iron Tablets (N=226)
Constipation (Gastrointestinal disorders) | 8 | 35
Diarrhea (Gastrointestinal disorders) | 8 | 13
Abdominal pain (Gastrointestinal disorders) | 12 | 6
Nausea (Gastrointestinal disorders) | 12 | 33
Fatigue (General disorders) | 13 | 5
Nasopharyngitis (Infections and infestations) | 7 | 14
Blood phosphorus decreased (Renal and urinary disorders) | 26 | 0
Headache (Nervous system disorders) | 34 | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less